CLINICAL TRIAL: NCT05090267
Title: Cognitive and Inflammation Targeted Gut-brain Interventions in Alcohol; Probiotics, Alcohol, Transcutaneous Vagus Nerve Stimulation, and HIV Study
Brief Title: The Path Study: Cognitive and Inflammation Targeted Gut-brain Interventions in Alcohol; Probiotics, Alcohol, Transcutaneous Vagus Nerve Stimulation, and HIV Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: University of Miami (Other); University of Louisville (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Exegi Pharma, LLC (Industry); Soterix Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: CED000000532; P01AA029543 (NIH); PRO00035889 (Other: UFIRST)
Record Dates: First submitted 2021-09-21; First posted 2021-10-22 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Cognition; Gut Microbiome

STUDY DESIGN:
Intervention Model Description: This is a 2 x 2 factorial, longitudinal design (tVNS/Sham, Probiotic/Placebo) across three time points (baseline; 30days and 90days).
Who Masked: Participant, Investigator
Masking Description: This is a 2x2 design in which subjects will be randomly assigned to one of 4 interventions groups: tVNS and probiotic (n=20); tVNS and placebo (n=20), sham stimulator and probiotic (n=20), and sham stimulator and placebo (n=20). We will use a computer-assisted stratified block randomization with block size of 4 to assign participants to the intervention. Study participants, investigators, staff, and physicians administering the probiotics or placebo will be unaware of specific group assignment. The stratified, blocked randomization and assignment of participants to the 4 intervention groups will be guided and monitored by Data Science Core.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Dietary Supplement (e.g., vitamins, minerals) (Experimental): Visbiome probiotic supplement
  Interventions: Dietary Supplement: Probiotic Supplement
- Device (including sham) (Active Comparator): Transcutaneous Vagal Nerve Stimulation (tVNS)
  Interventions: Device: Transcutaneous Vagal Nerve Stimulation (tVNS)

INTERVENTIONS:
Dietary Supplement: Probiotic Supplement — Participants will take a probiotic supplement or placebo for 90 days.
  Arms: Dietary Supplement (e.g., vitamins, minerals)
Device: Transcutaneous Vagal Nerve Stimulation (tVNS) — Participants will use a non-invasive stimulator 1 hour daily for 30 days. This stimulator is placed around the ear similar to headphones and produces a very mile electric current. This wellness device is safe to use and painless. Some describe the sensation to be a slight tingle up to a small itch.
  Arms: Device (including sham)

SUMMARY:
This project uses a hybrid trial design to evaluate two biomedical interventions targeting the gut-brain axis. One intervention is portable Transcutaneous Vagus Nerve Stimulator, tVNS, that is hypothesized to stimulate the autonomic nervous system, resulting in decreased inflammation and improved cognition. The second intervention is a probiotic supplement intended to replace gut bacteria that are associated with dysbiosis in persons with HIV and alcohol consumption.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-70 years
* English or Spanish speaking
* Alcohol users
* Cognitive impairment
* Current CD4>350

Exclusion Criteria:

* Diagnosed major psychiatric illness
* Consumption of over 300 drinks in the past 30 days
* Recent opioid use
* Lifetime history of medically-assisted alcohol detoxification
* Inpatient or intensive treatment for addictive behaviors in the past 12 months
* MRI contraindications
* Current antibiotic treatment
* Current probiotic use
* Physical impairment precluding motor response or lying still.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Improved cognition from day 1 to day 90 | Baseline up to 90 days
  Various indices of cognition will be measured using standard neuropsychological tests and neuroimaging at multiple time points and examined for change within subjects.
Reduction of dysbiosis from day 1 to day 90 | Baseline up to 90 days
  The gut microbiome will be analyzed through stool samples to measure for changes in biodiversity including an increase in beneficial bacteria.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Porges, PhD, Principal Investigator — University of Florida; Robert L Cook, MD, Study Director — University of Florida
Locations (1):
- University of Miami, Coral Gables, Florida, United States